CLINICAL TRIAL: NCT05700448
Title: A Phase III, Randomized, Double-Blind, Multicenter Study of Sugemalimab (CS1001) Plus PGemOx Regimen Versus Placebo Plus PGemOx for Subjects With Relapsed or Refractory Extranodal NK/T-Cell Lymphoma (R/R ENKTL)
Brief Title: Study of Sugemalimab (or Placebo) Plus PGemOx Regimen in Participants With Extranodal NK/T-Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS1001-306
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Extranodal NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — sugemalimab; pegaspargase; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugemalimab+PGemOx (Experimental): Participants receive sugemalimab 1200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) PLUS PGemOx regimen Q3W (pegaspargase 2000-2500 IU/m^2 via intramuscular injection on Day 1, gemcitabine 1000 mg/m^2 via IV infusion on Days 1 & 8 and oxaliplatin 130 mg/m^2 via IV infusion on Day 1.
  Interventions: Biological: Sugemalimab; Drug: Pegaspargase; Drug: Gemcitabine; Drug: Oxaliplatin
- Placebo+PGemOx (Placebo Comparator): Participants receive placebo via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) PLUS PGemOx regimen Q3W (pegaspargase 2000-2500 IU/m^2 via intramuscular injection on Day 1, gemcitabine 1000 mg/m^2 via IV infusion on Days 1 & 8 and oxaliplatin 130 mg/m^2 via IV infusion on Day 1.
  Interventions: Drug: Placebo; Drug: Pegaspargase; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Biological: Sugemalimab — IV infusion
  Arms: Sugemalimab+PGemOx
Drug: Placebo — IV infusion
  Arms: Placebo+PGemOx
Drug: Pegaspargase — Intramuscular injection
Drug: Gemcitabine — IV infusion
Drug: Oxaliplatin — IV infusion

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of sugemalimab (CS1001) in combination with PGemOx regimen (pegaspargase, gemcitabine, oxaliplatin) in treatment of adult patients with Extranodal NK/T-Cell Lymphoma (ENKTL) who have relapsed or become refractory to asparaginase-based regimens.

ELIGIBILITY:
Inclusion Criteria:

* Has ENKTL histologically confirmed by the study center. Nasal and non-nasal ENKTL are both allowed.
* Has relapsed or refractory ENKTL after prior asparaginase-based chemotherapy or chemoradiotherapy.
* Has Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
* Has at least one measurable lesion per Lugano 2014 classification.
* Is willing to provide stained tumor tissue sections and corresponding pathological reports or unstained tumor tissue sections (or tissue block) for central pathology review.
* Has adequate organ function.
* Has life expectancy of greater than 3 months.

Exclusion Criteria:

* Has aggressive natural killer-cell leukemia, current central nervous system (CNS) involvement or is concomitant with hemophagocytic lymphohistiocytosis.
* Has known additional malignancy within 5 years prior to randomization.
* Has an active autoimmune disease or has had an autoimmune disease that may relapse.
* Has had a major surgical procedure within 28 days or radiotherapy within 90 days before the first dose of study treatment.
* Has active tuberculosis infection.
* Has a known history of human immunodeficiency virus (HIV) infection and/or acquired immune deficiency syndrome (AIDS).
* Has a known active Hepatitis B or C virus infection.
* Has received systemic anti-cancer therapy within 28 days before the first dose of study treatment, including chemotherapy, immunotherapy, biological therapy (e.g. cancer vaccine, cytokine therapy or growth factors to treat cancer).
* Has used traditional Chinese medicines or herbal preparations with anti-tumor indications within 7 days before the first dose of study treatment.
* Has received systemic corticosteroid or any other immunosuppressive therapy within 14 days before the first dose of study treatment.
* Has received any treatment of antibody or drug that targets at T-cell coregulatory pathways or immune checkpoint pathways.
* Has toxicity from prior anti-cancer treatment, except for alopecia and fatigue, that has not recovered to baseline or ≤ Grade 1 according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0 before the first dose of study treatment.
* Has had allogenic hematopoietic stem cell transplantation (HSCT) within 5 years or autologous HSCT within 90 days before the first dose of study treatment.
* Has a known severe hypersensitivity to sugemalimab, its active substance and/or any of its excipients, or to other monoclonal antibodies.
* Female participants who are pregnant or breastfeeding.
* Is currently participating in or has participated in a trial of an investigational agent within 28 days before to the first dose of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) evaluated by blinded independent central review (BICR) according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification | Approximately 39 months after First Patient In

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately 39 months after First Patient In
Progression-free survival (PFS) evaluated by the Investigator according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification | Approximately 39 months after First Patient In
Objective response rate (ORR) evaluated by BICR and the Investigator according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification | Approximately 39 months after First Patient In
Duration of response (DoR) evaluated by BICR and the Investigator according to Criteria for Response Assessment of Lymphoma: Lugano 2014 Classification | Approximately 39 months after First Patient In

CONTACTS AND LOCATIONS:
Overall Officials: Qinzhou Qi, Study Director — CStone Pharmaceuticals